CLINICAL TRIAL: NCT02804087
Title: CALM-START - Controlling And Lowering Blood Pressure With the MobiusHDTM Device: STudying Effects in A Randomized Trial
Brief Title: Controlling And Lowering Blood Pressure With the MobiusHDTM Device
Acronym: CALM-START
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the rigorous nature of the trial and enrollment interruptions caused by COVID-19, the study enrolled only 4 of the planned 110 subjects. Due to the lack of enrollment, the study was closed.
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD0339
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MobiusHD Implantation (Experimental)
  Interventions: Device: MobiusHD
- Sham Implantation (Sham Comparator): Sham
  Interventions: Other: Sham Implantation

INTERVENTIONS:
Device: MobiusHD — The MobiusHD device is a self-expanding nitinol implant that is delivered intravascularly to the internal carotid sinus via the delivery catheter.
  Arms: MobiusHD Implantation
Other: Sham Implantation — Sham Implantation
  Arms: Sham Implantation

SUMMARY:
To evaluate the safety and performance of the MobiusHD system in subjects with resistant hypertension.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, sham-controlled, multi-center post market study investigating the efficacy and safety of MobiusHD System, and the efficacy of the MobiusHD device in lowering mean systolic 24-hour ABP in subjects with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years;
* Diagnosed with resistant hypertension;
* A mean systolic 24-hour ABP of 135-170 mmHg following at least 30 days on a stable antihypertensive medication regimen (no changes in medications or dose).
* A mean systolic 24-hour ABP of 135-170 mmHg after washout of all antihypertensive medications.

Exclusion Criteria:

* Known or clinically suspected baroreflex failure or autonomic neuropathy
* Treatable cause of resistant hypertension
* Hypertension secondary to an identifiable and treatable cause other than sleep apnea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
The change in mean systolic 24-hour ABP from baseline to 90 days post-randomization, between the treatment arm and the sham arm. | From Baseline to 90 days post-randomization
  Reduction in mean systolic 24-hour ABP

SECONDARY OUTCOMES:
Major adverse clinical events, including death, stroke, carotid interventions, and myocardial infarction, from baseline to 30 days post-randomization, between the treatment arm and the sham arm. | From Baseline to 30 days post-randomization
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Wilko Spiering, MD, Principal Investigator — UMC Utrecht; Jan Van der Heyden, MD, Principal Investigator — St. Antonius Hospital
Locations (4):
- Netherlands (4):
  - HagaZiekenhuis, The Hague, AA
  - Maastricht UMC+, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: No